CLINICAL TRIAL: NCT06824870
Title: Exploratory Study Evaluating the Effects of RV5026B Dermo-cosmetic Treatment ET1732 Formula Applied for 2 Months in Adult Subjects With Erythrocouperosis Associated With Pityriasis Folliculorum.
Brief Title: Exploratory Study Evaluating the Effects of Dermo-cosmetic RV5026B Applied for 2 Months in Adults With Erythrocouperosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV5026B20220514
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Erythrocouperose Associated With Pityriasis Folliculorum of the Face

STUDY DESIGN:
Intervention Model Description: During the first period, the tested product will be applied to the entire face.
  At Visit 2, after investigator assessments, the subjects will stop the study if they don't need a treatment by reference topical product. If they need it, they will continue the study and will apply:
  * the reference topical product, prescribed by the investigator on the entire face
  * the tested product on a single half-face according to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (first hemiface) (Experimental): Treated group = hemi-face with the reference topical product and the tested product RV5026B - ET1732 during period 2
- Control group (second hemiface) (Other): Control group = hemi-face with the reference topical product alone during period 2

INTERVENTIONS:
Other: RV5026B - ET1732 - Period 1 — Period 1 (1 month): The tested product RV5026B - ET1732 will be applied twice a-day on full-face The product sould be applied in sufficient quantity to cover the application area.
Drug: reference topical product - Period 2 — Period 2 (1 month) : the reference topical product, prescribed by the investigator will applied each evening on the whole face.
Other: RV5026B - ET1732 - Period 2 — Period 2 (1 month) : The tested product RV5026B - ET1732 will be applied twice a-day on randomised half-face. The evening application will be done 15 minutes after the application of the reference treatment. Hands must be washed between the application of the 2 products.

SUMMARY:
This exploratory study aims to evaluate the effects of the test product RV5026B - ET1732 on erythema, as well as on the sensations of discomfort and relief perceived in subjects with erythrocouperose and associated pityriasis folliculorum.

We wish to evaluate:

* firstly the test product alone in order to quantify the effects on the signs & symptoms on the entire face,
* then the contribution of the test product in addition to a reference topical treatment.

The test product RV5026B - ET1732 was developed to:

* Reduce redness, even if it has already set in, and help limit its reappearance
* Soothe the sensations of heating and discomfort associated

ELIGIBILITY:
Main inclusion criteria:

* Man or woman aged 18 to 75 years old
* Subject presenting erythrocouperosis associated with pityriasis folliculorum of the face with erythema of mild to severe intensity according to the IGA clinical rating on both cheeks
* High density of Demodex on both cheeks: SSSB1 > 5 D/cm² or SSSB2 > 10 D/cm²

Main non-inclusion criteria:

- Subject presenting, on the day of inclusion, a dermatological condition of the face other than that studied

1. ORAL/GENERAL TREATMENTS that were planned to be taken during the study OR that were taken:

   A. In the last 3 months:

   - Any change in hormone replacement therapy.

   - Any oral treatment Vit A or derivatives

   B. In the last 4 weeks:

   - Any change in oral drug treatment that could modify the skin characteristics of the subjects and interfere with the performance of the study product

   - Tetracyclines

   - Immunosuppressant

   - Antiparasitic

   - Corticosteroid or NSAID taken for more than 5 consecutive days

   C. In the last 2 weeks:

   - Antibiotic with known cutaneous impact
2. LOCAL TREATMENTS that were planned to be taken during the study OR that were taken:

   A. In the last 3 months:

   - Vascular laser of the face

   B. In the last 4 weeks:

   - Any topical medicinal product on the face that could modify the skin characteristics of the subjects and interfere with the performance of the study product.

   C. In the last 10 days:

   - Changes to any topical cosmetic product (toiletries, care products and makeup) on the face

   D. In the last 7 days:
   * Topical antiseptic on the face
   * Any topical cosmetic product applied to the face that could modify the skin characteristics of the subjects and interfere with the performance of the product under study

   E. Since the last wash performed the night before:

   - Application of topical treatment, rinsed or non-rinsed dermocosmetic product on the face

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Erythema score | Day 1, Day 29 & Day 57
  Assessed by the investigator according to the Investigator Global Assessment - IGA - scale (score from 0 to 3: None toSevere) on each side of the face
Overall dynamic efficiency score | Day 29 & Day 57
  Assessed by the investigator according to Investigator's Global Assessment (IGA) - (-3 to +3) (Very significant worsening = -3to Very significant improvement = +3) compared with baseline status at visit 1 on each side of the face
Demodex density | Day 1, Day 29 & Day 57
  assessed by Standardized Skin Surface Biopsy (SSSB1 & SSSB2 and SSSB1+2) on each hemiface by on-site optical microscope count, then protein analysis on SSSBs sample
Rating of the intensity of the erythema | Day 1, Day 29 & Day 57
  (score from 0 to 100) by centralized a posteriori analysis of the photographs taken on each side of the face, carried out by an expert dermatologist using software presenting the images taken for each of the subjects, blindly
Flush score | Day 1, Day 29 & Day 57
  Score over the last 3 days preceding the assessment according to the Global Flushing Severity Score - GFSS - numerical scale (score from 0 to 10 - None to Extreme: ) on each side of the face
Dynamic SGA (subject global assessment) scale | Day 1, Day 29 & Day 57
  Scale with 7 points (-3 to +3) (Very significant worsening = -3 to Very significant improvement = +3) in comparison with the initial state of visit 1 on each side
Subject acceptability questionnaire | Day 29 & Day 57
  assessed by the subject with subject's questionnaire
Tolerance of the products for 2 months of use by adverse events | Day 1, Day 29 & Day 57
  Recording of Adverse events
Tolerance of the tested product for 2 months of use by global tolerance per subject | Day 29 & Day 57
  assessed by the investigator for both groups and per subject, considering all individual AE and their characteristics, based on a 5-point scale (0=Bad tolerance, 4= Excellent tolerance)
Subject's compliance regarding the test product | During the entire course of the study (approximately 57 days)
  The subject will report his compliance in a subject's diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr FORTON, Schaarbeek, Belgium